CLINICAL TRIAL: NCT03472170
Title: Clinical Trial for Valuation of the Effectiveness of Lactoferrine in the Prevention of Sepsis in New Premature Born. Bimonitorization of the Antinflammatory Mechanisms, Antioxidants and the Intestinal Microbiote.
Acronym: LACTOPREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FCO-LAC-2016-01
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: SEPSIS SYNDROME
Keywords: bovine lactoferrin; late sepsis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): The nutritional supplement used will be bovine lactoferrin, a product marketed according to the regulations of the European Union, and approved by the European Food Safety Agency (EFSA) in 2012, and by the American Agency for Food and Drug Administration ( FDA) in 2013. It will be acquired after purchase from Dicofarm® (Rome, Italy).
  The Hospital Pharmacy Service will provide the established dose of lactoferrin, according to the administration schedule of 150 mg / kg / day (maximum 300 mg / day).
  The treatments will be administered in liquid form, in the least amount possible. The administration of lactoferrin will be carried out enterally, orally or by nasogastric tube.
  The intervention will be done in the first 72 hours of life, once a day, and for 4 weeks, extending to 6 weeks in the NB with EG ≤ 28 weeks and / or birth weight ≤ 1000 gr, or until discharge if this happens before.
  Interventions: Dietary Supplement: Enteral administration of bovine lactoferrin (bLf)
- Control Arm (Placebo Comparator): Placebo with similar visual and taste characteristics to the nutritional supplement of bovine lactoferrin.
  It will be administered in liquid form, in the least amount possible. The administration of placebo will be carried out enterally, orally or by nasogastric tube. The intervention will be done in the first 72 hours of life, once a day, and for 4 weeks, extending to 6 weeks in the NB with EG ≤ 28 weeks and / or birth weight ≤ 1000 gr, or until discharge if this happens before.
  Interventions: Other: Enteral administration of placebo

INTERVENTIONS:
Dietary Supplement: Enteral administration of bovine lactoferrin (bLf) — The pharmacy service of the hospital will provide the established dose of lactoferrin, according to the regimen of administration of 150 mg / kg / day (maximum 300 mg / day), as well as that of placebo. Both treatments will be administered in liquid form, in the least amount possible. Both the administration of lactoferrin and placebo will be carried out enterally, orally or by nasogastric tube. The intervention will be done in the first 72 hours of life, once a day, and for 4 weeks, extending to 6 weeks in the newborns with EG ≤ 28 weeks and / or birth weight ≤ 1000 gr, or until discharge if this happens before.
  Arms: Experimental Arm
Other: Enteral administration of placebo — Enteral administration of placebo with similar visual and gustatory characteristics in the first 72 hours of life, and for 4 weeks (6 weeks in the RN ≤ 1000 gr and / or EG ≤ 28 weeks).
  Arms: Control Arm

SUMMARY:
To evaluate the efficacy of enteral administration of bovine lactoferrin (bLf) in the reduction of probable late sepsis or microbiologically proven in preterm infants with birth weight ≤ 1500 gr and / or gestational age ≤ 32 weeks.

DETAILED DESCRIPTION:
To date there are no published clinical data that jointly assess the impact of direct Lf supplementation on oxidative status, on biomarkers of systemic inflammation and on the microbiota of premature infants with or without sepsis. Clarification of these additional questions is essential for a better understanding of the benefits and implications of enteral administration of Lf in preterm infants. The enteral administration of lactoferrin reduces the incidence of late sepsis in preterm infants of very low birth weight (BMPN). Enteral supplementation with lactoferrin in NBWNS can have a beneficial effect on the systemic oxidative and inflammatory state, and may contribute to the creation of a healthy faecal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Both groups will include male or female children born preterm with birth weight ≤ 1500 g and / or EG ≤ 32 weeks. All tutors of patients, must sign the informed consent.

Exclusion Criteria:

* In both groups those subjects who do not meet the age and weight established at birth, have> 72 hours of life at the time of inclusion, who do not sign informed consent or who have the following morbidities will be discarded: 1) Early sepsis or vertical; 2) Gastrointestinal congenital anomalies; 3) Chromosomopathies; 4) Congenital anomalies and / or genetic diseases without survival expectations; 5) Severe perinatal hypoxia.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of proven and probable late sepsis | 12 months
  To evaluate the efficacy of enteral administration of bovine lactoferrin (bLf) in the reduction of probable late sepsis or microbiologically proven in preterm infants with birth weight ≤ 1500 gr and / or gestational age ≤ 32 weeks.

SECONDARY OUTCOMES:
Perinatal history and demographic characteristics | At baseline.
  Description of the perinatal history and demographic characteristics in the subjects of two intervention groups (lactoferrin vs placebo).
Morbidities | From 72 hours until 4 weeks after birth
  Assess the possible differences between the two groups with respect to the following morbidities:
  Global mortality and / or attributable to late sepsis before hospital discharge
  * Necrotizing enterocolitis
  * Retinopathy of prematurity
  * Bronchopulmonary dysplasia
  * Cerebral hemorrhage and periventricular leukomalacia
  * Hospital stay
  * Seriousness of late sepsis
  * Food tolerance
Adverse effects | From 72 hours until 4 weeks after birth and in every visit (months 3, 6, 12 y 24 after hospital discharge).
  Evaluation of the safety of the administration of lactoferrin by monitoring possible adverse effects.
Parameters of inflammation and oxidative stress | 0-24 hours of life, 7-10 days, 14-17 days of life, and one last extraction at the end of treatment, at 28-31 days
  Biomonitoring parameters of inflammation and oxidative stress in both groups, comparing possible differences.
Intestinal microbiota | Before and after treatment
  Study and compare the composition of the intestinal microbiota between both groups. Its modification will be assessed before and after treatment, and the implication of its distortion in late sepsis.
Subgroups evaluation | At the end of the trial.
  Analyze the results based on subgroups established by gestational age, birth weight, type of feeding and etiology of sepsis.
Anthropometric parameters and neurodevelopment | At 2 years of corrected age
  Evaluation of anthropometric parameters and neurodevelopment at 2 years of corrected age.

CONTACTS AND LOCATIONS:
Overall Officials: María Dolores Ordoñez, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba
Locations (1):
- Hosìtal Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available.
  Individual parcicipant data that underlie the results reportes in this article, after deidenttification (text, tables, figures and appendices)
  The other documents that will be available: study protocol, Statistical Analysis Plan, Informed Consent Form.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Open under request.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.